CLINICAL TRIAL: NCT04331405
Title: Allogeneic Mononuclear Umbilical Cord Blood Systemic Infusions for Adult Patients With Severe Acute Contusion Spinal Cord Injury: Phase I Safety Study and Phase IIa Primary Efficiency Study
Brief Title: Allogeneic Cord Blood Cells for Adults With Severe Acute Contusion Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Collaborators: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Principal Investigator, Vladimir A. Smirnov, MD, Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41-18/03/2013
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Spinal Cord Contusion
Keywords: spinal cord injury; ASIA A/B; cell therapy; cord blood stem cells; regenerative medicine
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: 20 patients having acute contusion spinal cord injury (3 days post-trauma max) and ASIA A/B neurological deficit were divided into 2 groups: pilot group (n = 10) receiving hUCBMC treatment in addition to standard therapy and control group (n = 10) receiving standard treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot group (Experimental): 10 patients with acute severe contusion spinal cord injury (ASIA A/B) included into the group. Patients meeting inclusion/exclusion criteria underwent primary surgical treatment (decompression and stabilization) received hUCBMC infusions weekly (4 infusions overall) in addition to standard therapy during in-hospital treatment. After the discharge patients were examined for 4 times. Observation period was 1 year.
  Interventions: Biological: Human Allogeneic Umbilical Cord Blood Mononuclear Cells (hUCBMCs) systemic (i.v.) infusions
- Control group (No Intervention): 10 patients with acute severe contusion spinal cord injury (ASIA A/B) included into the group. Patients meeting inclusion/exclusion criteria underwent primary surgical treatment (decompression and stabilization) received standard therapy during in-hospital treatment. After the discharge patients were examined for 4 times. Observation period was 1 year.

INTERVENTIONS:
Biological: Human Allogeneic Umbilical Cord Blood Mononuclear Cells (hUCBMCs) systemic (i.v.) infusions — HUCBMCs samples were prepared for infusion in the specialized laboratory of Cord Blood Bank (CryoCenter Ltd) and transported to the clinic immediately within 2 hours in the Dry Shipper. All samples were chosen according to patients blood group and rhesus-factor.
  All samples were examined for hemotransmissive infections and cell viability prior to the preparation.
  Obtained samples were infused through the blood transfusion systems with additional filter after 3 tests for biological and individual compatibility and tolerance.
  Each patient of the pilot group received 4 cell infusions (1 infusion per week) with 1 week interval during the in-hospital treatment.
  Arms: Pilot group

SUMMARY:
Study evaluates the safety and primary efficiency of systemic (i.v.) allogeneic human umbilical cord blood mononuclear cell infusions in patients with severe acute contusion spinal cord injury (ASIA A/B). 20 patients were included. Half of patients received cell therapy in addition to standard therapy, while the other half received standard therapy only.

DETAILED DESCRIPTION:
Present study was prospective randomized open-label clinical study, Phases I/IIa. Randomization was performed using envelope method (50 envelopes including Cell Therapy and Standard Therapy, 25 of each).

20 patients with severe scute contusion spinal cord injury (cervical, thoracic and lumbar cone segments) were included into the study. Patients were divided into 2 groups: pilot group (n = 10) obtaining standard conservative therapy and 4 i.v. infusions of Human Allogeneic Umbilical Cord Blood Mononuclear Cells (hUCBMCs) (~ 300 M in 100 mL) and control group (n = 10) obtaining standard conservative therapy only. Cell Therapy was initiated in patients within 3 days after SCI episode after primary surgical decompression and/or stabilization was performed. Patients inclusion decision depended on meeting the inclusion/exclusion criteria and informed consent signed.

hUCBMC samples were prepared in the specialized laboratory and transported to the hospital immediately within 2 hours. Cells infusions were performed following 3 tests for biological compatibility and potential intolerance for each patient.

All four infusion were performed during in-hospital treatment. Observational period reached 1 year after SCI. All included patients were examined daily during in-hospital treatment following 4 times within observational period (1 year).

All adverse events and potential complications were analyzed within 1 year after SCI using CTCAE v5.0 classification.

Outcome parameters were analyzed at the end of observation and examined using standard statistical instruments.

ELIGIBILITY:
Inclusion Criteria:

* acute spinal cord injury (first 3 days after trauma)
* contusion type of SCI (MRI-confirmed)
* Russian citizenship
* Informed consent understood and signed by the patient

Exclusion Criteria:

* systolic arterial pressure (APsyst) > 185 mmHg OR diastolic AP (APdia) > 105 mmHg OR indications for aggressive AP lowering using i.v. therapy
* myocardial infarction within 3 months prior to SCI
* glucose level < 3.5 mM/L or > 21 mM/L
* organic CNS pathology
* acute internal organs diseases requiring surgical treatment
* autoimmune diseases
* serious surgical treatment or severe trauma within 3 months prior to SCI
* pregnancy or breast feeding
* acute infections including tuberculosis, syphilis, HIV, hepatitis B and C etc.
* severe acute and chronic hematological diseases
* rare patient's blood group parameters preventing adequate hUCBMCs sample selection (e.g. Kell+, A2B group, rare phenotype etc.)
* any benign or oncological tumors (if not fully treated prior to SCI)
* inability to participate in key examination following clinic discharge
* any psychiatric diseases preventing patient from informed consent OR treatment plan understanding
* confirmed hypersensitivity and/or allergy to any component of the studied biological compound
* inability to accomplish present study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 1 year
  All potential adverse events were analyzed during the first year after SCI. All adverse events (AEs) were classified using CTCAE v5.0 classification system in each of 10 patients of pilot group.
  Severity of AEs: Grade 1 - mild; asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2 - moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL; Grade 3 - severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; Grade 4 - life-threatening consequences; urgent intervention indicated; Grade 5 - death related to AE.
  Relationship to the investigated therapy method: Degree 1 - unrelated; Degree 2 - possibly related; Degree 3 - probably related; Degree 4 - definitely related.
Neurological Deficit Change [ASIA scale] | Change from Baseline at 1 year after SCI
  Dynamics of neurological deficit level within 1 year after SCI was analyzed using ASIA clinical scale: ASIA A - total motor and sensory impairment; ASIA B - total motor impairment and partial sensory impairment below SCI level or pelvic sensitivity preserved; ASIA C - incomplete motor (at least half of key muscle strength less than 3 points) and sensory impairment; ASIA D - incomplete motor (at least half of key muscle strength more than 3 points) and sensory impairment; ASIA E - normal. Neurological deficit level was compared between pilot and control groups.
Quality of Life [FIM scale] | 1 year after SCI
  Quality of life level was assessed within 1 year after SCI using FIM (functional impairment) scale. FIM scale evaluates 5 groups of parameters including motor functions and self-service, mobility, motion level, pelvic functions and intellectual functions (e.g. communication and social activity). Each group includes several parameters assessed using point system (maximum 7 points for each parameter). A total sum of points is counted and compared between pilot and control groups.

SECONDARY OUTCOMES:
Motor Deficit Change [Muscle Strength] | Change from Baseline at 1 year after SCI
  A dynamics of motor deficit was assessed using standard scale of key muscle strength. Two groups of parameters were considered including upper extremities strength (UEMS) and lower extremities strength (LEMS). Since patients with different SCI levels were included into the study (both cervical and thoracic/lumbar cone) LEMS parameter is more significant.
  Upper key muscles: C5 - biceps, С6 - wrist extensors, C7 - triceps, C8 - fingers flexors, Th1 - V finger abductor. Lower key muscles: L2 - m. psoas, L3 - quadriceps, L4 - m. tibialis anterior, L5 - I toe extensor, S1 - gastrocnemius.
  Both LEMS and cumulative (UEMS + LEMS) parameters were compared.
Independent Verticalization Ability | 1 year after SCI
  Patients ability to verticalize independently and mobility level were analyzed. First is determined by patient's ability to get up and stand more than 10 seconds without assistance. Second is determined by patient's ability to move without assistance depending on the distance: grade 1 - less than 10 m; grade 2 - less than 50 m; grade 3 - less than 100 m' grade 4 - 100 - 500 m; grade 5 - more than 500 m.
Lower Extremities Spasticity Level [Modified Asworth scale] | 1 year after SCI
  Spasticity level of lower extremities muscles was assessed using modified Ashworth scale. Grade 0 - no spasticity. Grade 1 - slight elevation of muscle tone, minimal tension at the end of movement amplitude during flexion and extension; Grade 1+ - slight elevation of muscle tone, minimal tension at least at half of movement amplitude. Grade 2 - moderate elevation of muscle tone during whole movement, but passive movements are not obstructed. Grade 3 - significant elevation of muscle tone, passive movements are partially obstructed. Grade 4 - rigid limb position in flexion or extension (contracture).
Feeling of Bladder Filling | 1 year after SCI
  Frequency of pelvic function disorders was assessed. Analysis included 2 parameters: (i) feeling of bladder filling and (ii) urinary inconsistence. First parameter is determined by patient's subjective feeling of bladder filling correlating to ultrasound confirmation of full bladder.
Urinary Inconsistence | 1 year after SCI
  Frequency of pelvic function disorders was assessed. Analysis included 2 parameters: (i) feeling of bladder filling and (ii) urinary inconsistence. Second parameter is determined by patient's ability for passive self-urination without application of any devices (e.g. urinary catheters, medical condoms or cystostomy).
Spinal Cord Conductivity [Electrophysiological assessment] | 1 year after SCI
  Spinal cord conductive function restoration was assessed using electrophysiological examination. Electroneuromyography supplemented with transcranial magnetic stimulation was performed to assess the level of signal conduction through the injured spinal cord. Significant diversity of SCI levels and baseline neurological deficit resulted in low significance of individual ENMG parameters comparison. Therefore only the parameters of conduction arrest was considered including (i) No conduction arrest (total or subtotal preservation of the overlay signal), (ii) Partial conduction arrest (decreased overlay signal) and (iii) Total conduction arrest (no overlay signal).

CONTACTS AND LOCATIONS:
Locations (1):
- N.V. Sklifosovsky Emergency Care Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
All the individual participant characteristics, assessed results of safety and efficiency evaluation, CT and MRI images can be provided to the interested persons and/or clinics via the contact with the Principal Investigator.